CLINICAL TRIAL: NCT00540644
Title: Phase II Study of Revlimid®, Oral Cyclophosphamide and Prednisone (RCP) for Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Phase II Study of Revlimid®, Oral Cyclophosphamide and Prednisone for Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Attaya Suvannasankha (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, Attaya Suvannasankha, Assistant Professor of Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0704-06; IUCRO-0170
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Revlimid
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Cyclophosphamide; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Revlimid, Cyclophosphamide, Prednisone (Experimental): Lenalidomide orally on Days 1-21 followed by 7 days rest, repeated every 28 days.
  Cyclophosphamide twice daily, orally on Days 1-21 followed by 7 days rest, repeated every 28 days.
  Prednisone every other day orally.
  Interventions: Drug: lenalidomide (Revlimid®); Drug: Cyclophosphamide; Drug: Prednisone

INTERVENTIONS:
Drug: lenalidomide (Revlimid®) — 25 mg p.o. daily on days 1-21 of each 28 day cycle
  Other Names: Revlimid®
Drug: Cyclophosphamide — 50 mg p.o. BID daily on days 1-21 of each 28 day cycle
Drug: Prednisone — 50 mg p.o. Q.O.D.

SUMMARY:
The purpose of this study to explore the combination of Revlimid®, oral cyclophosphamide and prednisone (RCP) in patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
This is a phase II single institution trial in patients with newly diagnosed multiple myeloma. Revlimid® 25 mg p.o. daily on days 1-21 of each 28-day cycle. Cyclophosphamide 50 mg p.o. BID daily on days 1-21 of each 28-day cycle. Prednisone 50 mg p.o. Q.O.D..

ELIGIBILITY:
Inclusion Criteria:

Patients with newly diagnosed, symptomatic multiple myeloma based on the following criteria:

* Presence of an M-component in serum and/or urine plus clonal plasma cells in the bone marrow and/or a documented clonal plasmacytoma

PLUS one or more of the following:

* Calcium elevation (11.5 mg/dl) [42.65 mmol/l]
* Renal insufficiency (1.5 x the ULN of serum creatinine)
* Anemia (hemoglobin <=10 g/dl or 2 g/dl <= normal)
* Bone disease (lytic lesions or osteopenia)

Measurable disease is defined at least one of the following three measurements:

* Serum M-protein >=1 g/dl ( or 10 g/l)
* Urine M-protein >=200 mg/24 h
* Serum FLC assay: Involved FLC level >=10 mg/dl (>=100 mg/l) provided serum FLC ratio is abnormal
* Measurable plasmacytoma
* NOTE: If a patient meets the criteria for symptomatic multiple myeloma but does not meet serum M-protein, urine M-protein or serum FLC levels stated above, percent plasma cells in bone marrow will be used to follow response.

Laboratory test results within these ranges:

* Absolute neutrophil count >= 1.0 x 109/L
* Platelet count >= 50 x 10(9)/L
* Hemoglobin >= 9 gm/dl
* Serum creatinine <= 2.5mg/dL.
* Total bilirubin <=1.5 x upper limit of normal
* AST (SGOT) and ALT (SGPT) <= 3 x ULN

Exclusion Criteria:

* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Patients with a solitary plasmacytoma
* Patients with uncontrolled diabetes
* Patients with ≥ Grade 3 sensory neuropathy
* History of cardiac disease, with NYHA Class II or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Attaya Suvannasankha, M.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Original Study - Revlimid, Cyclophosphamide, Prednisone: Original portion of the study where patients received Revlimid® 25 mg p.o. daily on days 1-21 of each 28-day cycle. Cyclophosphamide 50 mg p.o. BID daily on days 1-21 of each 28-day cycle. Prednisone 50 mg p.o. Q.O.D.
- Extension - Revlimid, Cyclophosphamide, Prednisone: Extension portion of the study where patients received Revlimid® 25 mg p.o. daily on days 1-21 of each 28-day cycle. Cyclophosphamide 50 mg p.o. BID daily on days 1-21 of each 28-day cycle. Prednisone 50 mg p.o. Q.O.D.
Period: Overall Study
Arm/Group | Original Study - Revlimid, Cyclophosphamide, Prednisone | Extension - Revlimid, Cyclophosphamide, Prednisone
Started | 48 | 22
Completed | 39 | 13
Not Completed | 9 | 9
Not completed — Adverse Event | 3 | 1
Not completed — Disease Progression | 3 | 1
Not completed — Physician Decision | 0 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Noncomplilance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Original Study - Revlimid, Cyclophosphamide, Prednisone | Extension - Revlimid, Cyclophosphamide, Prednisone | Total
Number analyzed (Participants) | 48 | 22 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 17 | 43
  >=65 years | 22 | 5 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10.5) | 59.9 (8.0) | 61.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 8 | 26
  Male | 30 | 14 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 48 | 22 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 43 | 21 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR) After 6 Cycles of Therapy Using the Proposed International Myeloma Working Group Uniform Response Criteria
Description: Evaluate the response rate of patients receiving therapy. Patients are considered as having a response if their overall response is Partial Response or better using the proposed International Myeloma Working Group uniform response criteria. The percentage of patients achieving this and the exact 95% confidence interval will be calculated.
Time Frame: After 6 cycles
Population: All patients receiving at least one dose of study drug and having at least one post-baseline visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Original Study - Revlimid, Cyclophosphamide, Prednisone | Extension - Revlimid, Cyclophosphamide, Prednisone
Number analyzed (Participants) | 45 | 21
percentage of participants | 86.7 [73.2 to 95.0] | 71.4 [47.8 to 88.7]

2. Secondary Outcome: Treatment Related Adverse Events Grade 3 or Higher
Description: Number of unique patients who had treatment related (possible, probable or definite) adverse events that were graded 3 or greater.
Time Frame: Beginning of treatment up to 5 years
Population: All patients enrolled and received treatment.
Measure: Number; unit: participants
Arm/Group | Original Study - Revlimid, Cyclophosphamide, Prednisone | Extension - Revlimid, Cyclophosphamide, Prednisone
Number analyzed (Participants) | 48 | 22
participants | 21 | 11

3. Secondary Outcome: Quality of Life Using the FACT-G Data
Description: Change from baseline FACT-G scores. The quality of life questionnaire (FACT-G) was given at various timepoints during the study. The values for change from baseline to endpoint are provided.
  Physical Well-Being (PWB; sum of 7 items, point range 0-28); Social/Family Well-Being (SWB, sum of 7-items, point range 0-28); Emotional Well-Being (EWB; sum of 6-items, point range 0-24); Functional Well-Being (FWB; sum of 7-items, point range 0-28) ; Fact-G score=sum of PWB, SWB, EWB, FWB, point range 0-108. Note: The higher the score, the better the outcome
Time Frame: baseline and after last cycle (up to 6 cycles)
Population: All patients enrolled and received treatment with a baseline and post-baseline measurement.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Original Study - Revlimid, Cyclophosphamide, Prednisone | Extension - Revlimid, Cyclophosphamide, Prednisone
Number analyzed (Participants) | 29 | 15
scores on a scale
  Physical Well-Being Change from Baseline | 1.57 (6.20) | -2.81 (6.14)
  Social/Family Well-Being Change from Baseline | -0.03 (5.08) | -0.23 (3.53)
  Emotional Well-Beling Change from Baseline | 2.52 (3.95) | 0.60 (3.22)
  Functional Well-Being Change from Baseline | 3.38 (5.33) | -1.17 (4.97)
  FACT-G Change from Baseline | 7.44 (13.07) | -3.61 (10.92)

ADVERSE EVENTS:
Time Frame: up to 5 years
Arm/Group | Original Study - Revlimid, Cyclophosphamide, Prednisone | Extension - Revlimid, Cyclophosphamide, Prednisone
Serious Adverse Events (participants affected / at risk) | 12/48 | 5/22
Other Adverse Events (participants affected / at risk) | 48/48 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Original Study - Revlimid, Cyclophosphamide, Prednisone (N=48) | Extension - Revlimid, Cyclophosphamide, Prednisone (N=22)
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (Blood and lymphatic system disorders) | 2 | 1
CARDIAC GENERAL - OTHER (Cardiac disorders) | 1 | 0
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2 | 0
INFECTION (DOCUMENTED CLINICALLY OR MICROBIOLOGICALLY) WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E (Infections and infestations) | 1 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - LUNG (PNEUMONIA) (Infections and infestations) | 1 | 0
HEMOGLOBIN (Investigations) | 0 | 1
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Investigations) | 1 | 1
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 1 | 2
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 1 | 0
SEIZURE (Nervous system disorders) | 1 | 0
CONFUSION (Psychiatric disorders) | 1 | 1
RENAL FAILURE (Renal and urinary disorders) | 2 | 1
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
FLU-LIKE SYNDROME (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Original Study - Revlimid, Cyclophosphamide, Prednisone (N=48) | Extension - Revlimid, Cyclophosphamide, Prednisone (N=22)
PALPITATIONS (Cardiac disorders) | 2 | 1
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - SINUS BRADYCARDIA (Cardiac disorders) | 0 | 1
AUDITORY/EAR - OTHER (Ear and labyrinth disorders) | 0 | 1
OTITIS, MIDDLE EAR (NON-INFECTIOUS) (Ear and labyrinth disorders) | 0 | 1
OCULAR/VISUAL - OTHER (Eye disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 15 | 9
DIARRHEA (Gastrointestinal disorders) | 13 | 12
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 | 1
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 1 | 1
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 1 | 3
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 9 | 6
HEMORRHOIDS (Gastrointestinal disorders) | 0 | 2
NAUSEA (Gastrointestinal disorders) | 14 | 8
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 5 | 3
PAIN - PELVIS (Gastrointestinal disorders) | 0 | 2
VOMITING (Gastrointestinal disorders) | 3 | 2
EDEMA: LIMB (General disorders) | 14 | 8
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 24 | 14
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 5 | 7
PAIN - CHEST/THORAX NOS (General disorders) | 4 | 2
PAIN - FACE (General disorders) | 0 | 1
PAIN - OTHER (General disorders) | 6 | 5
RIGORS/CHILLS (General disorders) | 6 | 4
INFECTION (DOCUMENTED CLINICALLY OR MICROBIOLOGICALLY) WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E (Infections and infestations) | 2 | 3
INFECTION - OTHER (Infections and infestations) | 1 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - BLADDER (URINARY) (Infections and infestations) | 1 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - DENTAL-TOOTH (Infections and infestations) | 1 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - LUNG (PNEUMONIA) (Infections and infestations) | 2 | 1
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - UPPER AIRWAY NOS (Infections and infestations) | 3 | 2
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - URINARY TRACT NOS (Infections and infestations) | 1 | 1
INFECTION WITH UNKNOWN ANC - LUNG (PNEUMONIA) (Infections and infestations) | 0 | 1
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Injury, poisoning and procedural complications) | 0 | 2
BURN (Injury, poisoning and procedural complications) | 0 | 1
FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTEREMIA) (Investigations) | 0 | 1
CREATININE (Investigations) | 0 | 1
HEARING: PATIENTS WITH/WITHOUT BASELINE AUDIOGRAM AND ENROLLED IN A MONITORING PROGRAM (Investigations) | 0 | 1
HEMOGLOBIN (Investigations) | 2 | 1
METABOLIC/LABORATORY - OTHER (Investigations) | 1 | 1
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Investigations) | 7 | 6
PLATELETS (Investigations) | 3 | 0
ANOREXIA (Metabolism and nutrition disorders) | 6 | 6
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 1
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Metabolism and nutrition disorders) | 1 | 1
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTRAOCULAR (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 5 | 1
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTREMITY-UPPER (Musculoskeletal and connective tissue disorders) | 5 | 1
MUSCULOSKELETAL/SOFT TISSUE - OTHER (Musculoskeletal and connective tissue disorders) | 3 | 3
OSTEONECROSIS (AVASCULAR NECROSIS) (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 19 | 9
PAIN - BONE (Musculoskeletal and connective tissue disorders) | 12 | 7
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 6 | 5
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 14 | 5
PAIN - MUSCLE (Musculoskeletal and connective tissue disorders) | 2 | 3
PAIN - NECK (Musculoskeletal and connective tissue disorders) | 2 | 2
ATAXIA (INCOORDINATION) (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 9 | 4
NEUROPATHY: SENSORY (Nervous system disorders) | 13 | 6
PAIN - HEAD/HEADACHE (Nervous system disorders) | 2 | 2
PAIN - SINUS (Nervous system disorders) | 0 | 1
SOMNOLENCE/DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
SYNCOPE (FAINTING) (Nervous system disorders) | 3 | 1
TASTE ALTERATION (DYSGEUSIA) (Nervous system disorders) | 2 | 2
TREMOR (Nervous system disorders) | 7 | 3
INSOMNIA (Psychiatric disorders) | 18 | 7
MOOD ALTERATION - ANXIETY (Psychiatric disorders) | 4 | 2
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 2 | 2
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 0 | 2
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 2 | 1
VAGINAL DRYNESS (Reproductive system and breast disorders) | 0 | 1
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Respiratory, thoracic and mediastinal disorders) | 2 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 | 5
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 10 | 12
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - NOSE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PAIN - THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 3 | 3
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 2 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 3
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 16 | 2
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 16 | 8
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 4 | 1
SWEATING (DIAPHORESIS) (Skin and subcutaneous tissue disorders) | 10 | 6
HYPERTENSION (Vascular disorders) | 1 | 1
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes